CLINICAL TRIAL: NCT05626972
Title: A Multi-center, Randomized, Open-label Blinded Endpoint (PROBE), Phase III Study, for the Comparation of Tenecteplase (TNK) Versus Alteplase, With a 1:1 Allocation, Before Thrombectomy in Patients With Acute Ischemic Stroke and Large Vessel Occlusion Suspicion in Catalonia (TNK-CAT)
Brief Title: Tenecteplase Compared to Alteplase for Patients With Large Vesel Oclusion Suspicion Before Thrombectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-001599-13
Record Dates: First submitted 2022-11-04; First posted 2022-11-25 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; large vessel occlusion
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Clinical outcome at day 90 will be obtained by centralized telephone call of the mRS in a blinded manner by certified personnel of the Catalan Stroke Program.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenecteplase (TNK) (Active Comparator): Drug: Alteplase (tPA) Dose: 0.9 mg/kg Route: Intravenous (IV) infusion
  Interventions: Drug: Tenecteplase
- Alteplase (tPA) (Active Comparator): Drug: Tenecteplase (TNK) Dose: 0.25 mg/kg Route: Intravenous (IV) bolus injection
  Interventions: Drug: Tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Patients will be randomized 1:1 to standard dose tPA (0.9 mg/kg) or TNK (0.25mg/kg) before endovascular therapy (EVT)

SUMMARY:
Background: The TNKCAT trial represents an innovative approach to optimize timely reperfusion in the Mothership and Drip-and-Ship scenarios. The logistic advantage of a single bolus infusion of TNK (compared to 1-h infusion of tPA) would markedly reduce the needle-to-groin and Door-in- door-out time. The implementation of a quality improvement package (QIP) in the TNKCAT trial would directly improve the quality and efficiency of the Health Care System. In addition, an improvement of transfer models would reduce the cost of unnecessary transfers, together with the fact that TNK is up to 50% less expensive than tPA, makes the TNKCAT in firm line with the sustainability strategy of the National Health Care system.

Outcomes: The aim of the present study is to determine the safety and efficacy of TNK (0.25mh/kg) compared to tPA (0.9 mg/kg) in patients with Large Vessel Occlusion (LVO) suspicion, candidates for thrombectomy, in both Mothership and Drip-and-Ship scenarios.

Study Duration: 2 years. Patients will participate in the trial for 3 months.

Study design: Multicentre, prospective, randomized open-label blinded endpoint (PROBE) phase III study in acute stroke patients with LVO suspicion within 4.5 hours of stroke onset, candidates for EVT. Patients will be randomized 1:1 to standard dose tPA (0.9 mg/kg) or TNK (0.25mg/kg) before EVT.

Clinical, imaging and outcome data will be collected at baseline, 24-36 hours, day 3, day 5 and day 90.

Estimated enrollment: 500 patients

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible to undergo intravenous thrombolysis (tPA or TNK) within 4.5 hours after the onset of ischemic stroke.
* Suspicion of Cerebral vascular occlusion on brain imaging.
* Age >18 years old
* Men and women (women with child-bearing potential are excluded, unless pregnancy test negative/ confirmed menstrual period/ postmenopausal or hysterectomy).
* A new focal disabling neurologic deficit consistent with acute cerebral ischemia.
* Informed consent obtained from subject or acceptable subject surrogate (i.e. next of kin, or legal representative), or Differed Inform Consent (DIC) to avoid any delay in the initiation of iv thrombolysis. The DIC will be sign by the patient or next of kin at any time after the tPA or TNK treatment is started.

Exclusion criteria:

* Patients with severe preexisting disability, defined as a modified Rankin scale score >3.
* Glasgow Coma Scale score ≤ 7.
* Known hemorrhagic diathesis, coagulation factor deficiency, or antivitamin K oral anticoagulant therapy with INR >3.0. Subjects on factor Xa inhibitors (e.g. apixaban) or direct thrombin inhibitors are eligible for participation.
* Severe, sustained and uncontrollable hypertension (systolic blood pressure >185 mmHg or diastolic blood pressure >110 mmHg).
* Serious, advanced, or terminal illness with anticipated life expectancy of less than 3 months.
* Patients that are unlikely to be available for a 90-day follow-up (e.g. no fixed home address, visitor from overseas).
* Patient participating in a randomized study, involving an investigational drug or device that would impact this study.
* Suspicion of aortic dissection presumed septic embolus, or suspicion of bacterial endocarditis.

Imaging exclusion criteria:

* Clinical symptoms suggestive of bilateral stroke or stroke in multiple territories.
* Cerebral vasculitis.
* CT or MRI evidence of hemorrhage
* Significant mass effect with midline shift.
* Evidence of intracranial tumor.
* Subjects with known occlusions in multiple vascular territories (e.g., bilateral anterior circulation, or anterior/posterior circulation).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin scale score at 3 months | 3 months
  Shift analysis of the modified Rankin scale score at 3 months
Mortality rate | 3 months
  Mortality at 3 months
Symptomatic intracerebral haemorrhage (ICH) and neurological deterioration | 24 -36hours
  Symptomatic ICH defined as intracerebral haemorrhage (PH2) within 36 hours of treatment, combined with neurological deterioration leading to an increase of ≥ 4 points on the National institute of Health Stroke Scale (NIHSS) from baseline, or the lowest NIHSS value between baseline and 24 hours.

SECONDARY OUTCOMES:
Rates of mRS 0-1 at 3 months | 3 months
  Modified Rankin scale score (0-1) rates
Rates of mRS 0-2 at 3 months | 3 months
  Modified Rankin scale score (0-2) rates
Rates of pre-interventional recanalization | during the procedure
  Recanalization rate
Dramatic clinical recovery before endovascular treatment (EVT) | before the procedure
  Dramatic clinical recovery before EVT (Improvement in > 8 points in the NIHSS score or NIHSS score < 2 before groin puncture)
First pass TICI 3, final TICI 2b-3 | immediately after the procedure
  Rates of first pass TICI 3, final TICI 2b-3
Distal embolization during EVT | during the procedure
  Rates of distal embolization during EVT
Needle-to-groin times and DIDO times | immediately after the procedure
  Differences in needle-to-groin times in Mothership patients and in DIDO times in Drip-and-Ship patients.
Time metrics between TNKCAT and non-TNKCAT centers | at the end of the study
  Differences in time metrics between TNKCAT and non-TNKCAT centers
Final infarct volume on follow up CT | 24-36 hours follow up
  Differences in final infarct volume on follow up CT

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No